CLINICAL TRIAL: NCT07060807
Title: An Open-label, Randomized, Phase 3 Study to Evaluate Patritumab Deruxtecan Monotherapy Versus Treatment of Physician's Choice in Hormone Receptor-positive, HER2-negative Unresectable Locally Advanced or Metastatic Breast Cancer (HERTHENA-Breast04)
Brief Title: A Clinical Study of Patritumab Deruxtecan to Treat Breast Cancer (MK-1022-016)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1022-016; U1111-1317-5490 (Registry Identifier: UTN); 2025-520582-51-00 (Registry Identifier: EU CT); jRCT2031250297 (Registry Identifier: Japan Registry of Clinical Trial (jRCT))
Record Dates: First submitted 2025-07-02; First posted 2025-07-11 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — patritumab deruxtecan; Paclitaxel; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Capecitabine; liposomal doxorubicin; trastuzumab deruxtecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Patritumab Deruxtecan (Experimental): Participants receive patritumab deruxtecan via intravenous (IV) infusion every 3 weeks (Q3W) for approximately 13 months.
  Interventions: Biological: Patritumab deruxtecan
- Treatment of Physician's Choice (Active Comparator): Participants receive treatment of physician's choice (TPC) for up to 13 months. The TPC may be any of the following options: Paclitaxel (80 mg/m^2) on Days 1, 8, 15, and 22 of each 4-week cycle; Paclitaxel (90 mg/m^2) on Days 1, 8, and 15 of each 4-week cycle; Nab-paclitaxel (100 mg/m^2) on Days 1, 8, and 15 of each 4-week cycle; Capecitabine (1000 mg/m^2) bid on Days 1 to 14 of each 3-week cycle; Liposomal doxorubicin (50 mg/m^2) on Day 1 of each 4-week cycle; or trastuzumab deruxtecan (T-DXd) (5.4 mg/kg) Q3W.
  Interventions: Drug: Paclitaxel; Drug: Nab-paclitaxel; Drug: Capecitabine; Drug: Liposomal doxorubicin; Biological: Trastuzumab deruxtecan

INTERVENTIONS:
Biological: Patritumab deruxtecan — Administered via intravenous (IV) infusion
  Other Names: MK-1022; HER3-DXd; U3-1402
  Arms: Patritumab Deruxtecan
Drug: Paclitaxel — Administered via IV infusion
  Other Names: TAXOL®; ONXAL®
  Arms: Treatment of Physician's Choice
Drug: Nab-paclitaxel — Administered via IV infusion
  Other Names: Abraxane®
  Arms: Treatment of Physician's Choice
Drug: Capecitabine — Administered via oral tablets
  Other Names: XELODA®
  Arms: Treatment of Physician's Choice
Drug: Liposomal doxorubicin — Administered via IV infusion
  Other Names: Doxil®
  Arms: Treatment of Physician's Choice
Biological: Trastuzumab deruxtecan — Administered via IV infusion
  Other Names: T-DXd; Enhertu®
  Arms: Treatment of Physician's Choice

SUMMARY:
Researchers are looking for other ways to treat breast cancer (BC) that is hormone receptor-positive and human epidermal growth factor receptor 2-negative (HR+/HER2-) and either unresectable locally advanced or metastatic.

* HR positive (HR+) means the cancer cells have proteins that attach to estrogen or progesterone (hormones) which help the cancer to grow and spread
* HER2 negative (HER2-) means the cancer cells have a low amount of a protein called HER2
* Unresectable locally advanced means the cancer cannot be completely removed by surgery and has spread into nearby tissue or muscles
* Metastatic means the cancer has spread to other parts of the body

Treatment for this type of breast cancer usually includes endocrine therapy (ET) and sometimes a second treatment. The main goal of this study is to learn if people who receive patritumab deruxtecan (also known as HER3-DXd and MK-1022) live longer overall or without the cancer growing/spreading, compared to people who receive chemotherapy or a different drug called trastuzumab deruxtecan.

ELIGIBILITY:
Inclusion Criteria:

The main inclusion criteria include but are not limited to the following:

* Has a diagnosis of hormone receptor positive (HR+)/human epidermal growth factor receptor 2 (HER2)- invasive breast carcinoma that is either locally advanced disease not amenable to resection with curative intent (herein called unresectable) or metastatic disease not treatable with curative intent
* Has centrally-confirmed HR+ and HER2- results and human epidermal growth factor receptor 3 (HER3) evaluable results from a biopsy obtained from a distant metastatic site or a locally advanced lesion on or after the most recent line of therapy (with certain exceptions)
* Must have had progression or recurrence on prior cyclin-dependent kinase (CDK)4/6 inhibitor + endocrine therapy (ET) with one of the following:

  * Radiographic disease progression, as assessed by the investigator, on CDK4/6 inhibitor + ET as 1L for treatment of unresectable locally advanced or metastatic HR+/HER2- breast cancer. CDK4/6 inhibitor + ET must be the only line of therapy received in the advanced setting, or
  * Disease recurrence, either radiographic and/or confirmed histologically via biopsy as assessed by the investigator, while on adjuvant ET in combination with a CDK4/6 inhibitor OR within 24 months from the date of last dose of adjuvant CDK4/6 inhibitor
* Has measurable disease per RECIST 1.1 as assessed by the local site investigator/radiology
* Human immunodeficiency virus (HIV)-infected participants must have well controlled HIV on antiretroviral therapy
* Has an Eastern Cooperative Oncology Group performance status of 0 or 1 assessed within 7 days before randomization

Exclusion Criteria:

The main exclusion criteria include but are not limited to the following:

* Has breast cancer amenable to treatment with curative intent
* Is eligible to receive additional endocrine-based treatment in the advanced setting as determined by the investigator
* Has a known germline breast cancer gene (BRCA) mutation (deleterious or suspected deleterious) where poly (ADP-ribose) polymerase (PARP) inhibitor(s) is a potential treatment option
* Has current visceral crisis or is at risk for impending visceral crisis that has or may cause imminent organ compromise and/or other life-threatening complications
* Has any of the following: a pulse oximeter reading <92% at rest, or requires intermittent supplemental oxygen, or requires chronic supplemental oxygen
* Has uncontrolled, significant cardiovascular disease or cerebrovascular disease
* Has ≥Grade 2 peripheral neuropathy.
* Has clinically significant corneal disease
* Has received prior chemotherapy for unresectable locally advanced or metastatic breast cancer
* Has received prior treatment with an anti-HER3 antibody and/or antibody-drug conjugate that consists of a topoisomerase I inhibitor (eg, T-DXd) or any other topoisomerase I inhibitor therapy
* Has received prior systemic anticancer therapy within 4 weeks (or 5 half-lives, whichever is shorter) before randomization; participants previously treated with ET plus a CDK4/6 inhibitor may participate as long as at least 2 weeks have elapsed since the last dose of therapy was administered
* Has received prior radiotherapy for non-central nervous system disease, or required corticosteroids for radiation-related toxicities, within 14 days of the first dose of study intervention
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has known additional malignancy that is progressing or has required active treatment within the past 3 years
* Has history of (noninfectious) pneumonitis/interstitial lung disease (ILD) that required steroids, has current pneumonitis/interstitial lung disease, or has suspected ILD/pneumonitis that cannot be ruled out by imaging at Screening
* Has severe hypersensitivity (≥Grade 3) to HER3-DXd and/or any of its excipients
* Has severe hypersensitivity (≥Grade 3) to all the available TPC and/or any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-21 (Actual); Primary Completion 2033-07-14 (Estimated); Study Completion 2033-07-14 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | Up to approximately 45 months
  PFS is defined as the time from first day of study intervention to the first documented progressive disease (PD) or death due to any cause, whichever occurs first as assessed by blinded independent central review (BICR). Per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions is also considered PD. The appearance of one or more new lesions is also considered PD. PFS as assessed by BICR will be presented.
Overall Survival (OS) | Up to approximately 85 months
  OS is the length of time from when the participant starts treatment until death from any cause.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to approximately 85 months
  ORR is defined as the percentage of participants with Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by BICR.
Duration of Response (DOR) | Up to approximately 85 months
  For participants who demonstrate a confirmed Complete Response (CR: disappearance of all target lesions) or Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1, DOR is defined as the time from first documented evidence of CR or PR until progressive disease (PD) or death. Per RECIST 1.1, PD is defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered PD. DOR as assessed by BICR will be presented.
Change from Baseline in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better outcome. The change from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score (the standardized average of the raw scores) will be presented.
Change from Baseline in the EORTC-QLQ-C30 Physical Functioning (Items 1-5) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate better physical functioning. The change from baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) combined score (the standardized average of the raw scores) will be presented.
Change from Baseline in the EORTC-QLQ-C30 Emotional Functioning (Items 1-5) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. Participant responses to 4 questions about their emotional functioning (Items 21-24) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate better emotional functioning. The change from baseline in EORTC QLQ-C30 Emotional Functioning (Items 21-24) combined score (the standardized average of the raw scores) will be presented.
Change from Baseline in the EORTC-QLQ-C30 Pain (Items 9 and 19) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. Participant responses to 2 questions about their pain (Items 9 and 19) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate greater pain. The change from baseline in EORTC QLQ-C30 Pain (Items 9 and 19) combined score (the standardized average of the raw scores) will be presented.
Time to First Deterioration (TTD) in the European Organization for Research and Treatment of Cancer (EORTC)-Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status (Item 29) and Quality of Life (Item 30) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of life (QoL) questionnaire. Participant responses to the questions regarding Global Health Status (GHS; "How would you rate your overall health during the past week?") and Quality of Life (QoL; "How would you rate your overall quality of life during the past week?") are scored on a 7-point scale (1= Very poor to 7=Excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better outcome. The TTD from baseline in GHS (EORTC QLQ-C30 Item 29) and QoL (EORTC QLQ-C30 Item 30) combined score (the standardized average of the raw scores), defined as the time from baseline to the first onset of a 10 or more points deterioration from baseline, will be presented.
TTD in the EORTC-QLQ-C30 Physical Functioning (Items 1-5) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. Participant responses to 5 questions about their physical functioning (Items 1-5) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate better physical functioning. The TTD from baseline in EORTC QLQ-C30 Physical Functioning (Items 1-5) combined score (the standardized average of the raw scores), defined as the time from baseline to the first onset of a 10 or more points deterioration from baseline, will be presented.
TTD in the EORTC-QLQ-C30 Emotional Functioning (Items 1-5) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. Participant responses to 4 questions about their emotional functioning (Items 21-24) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate better emotional functioning. The TTD from baseline in EORTC QLQ-C30 Emotional Functioning (Items 21-24) combined score (the standardized average of the raw scores) defined as the time from baseline to the first onset of a 10 or more points deterioration from baseline, will be presented.
TTD in the EORTC-QLQ-C30 Pain (Items 9 and 19) Combined Score | Baseline and up to approximately 85 months
  The EORTC QLQ-C30 is a cancer specific health-related quality-of-life questionnaire. Participant responses to 2 questions about their pain (Items 9 and 19) are scored on a 4-point scale (1=Not at All to 4=Very Much). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. Higher scores indicate greater pain. The TTD from baseline in EORTC QLQ-C30 Pain (Items 9 and 19) combined score (the standardized average of the raw scores), will be presented.
Number of Participants Who Experience One or More Adverse Event (AEs) | Up to approximately 85 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinue Study Treatment Due to an AE | Up to approximately 85 months
  An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a preexisting condition that is temporally associated with the use of the Sponsor's product, is also an AE. The number of participants who discontinue study treatment due to an AE will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (122):
- United States (25):
  - Southern Cancer Center (SCC) ( Site 8000), Daphne, Alabama
  - Los Angeles Hematology Oncology Medical Group ( Site 0026), Los Angeles, California
  - Hoag Memorial Hospital Presbyterian ( Site 0025), Newport Beach, California
  - St. Marys Hospital and Regional Medical Center-SCL Health Cancer Centers of Colorado ( Site 0021), Grand Junction, Colorado
  - Comprehensive Hematology Oncology ( Site 0060), St. Petersburg, Florida
  - Baptist Health Lexington ( Site 0050), Lexington, Kentucky
  - Baptist Health Hamburg ( Site 0071), Lexington, Kentucky
  - Rutgers Cancer Institute of New Jersey ( Site 0033), New Brunswick, New Jersey
  - Presbyterian Kaseman Hospital ( Site 0072), Albuquerque, New Mexico
  - University of New Mexico Comprehensive Cancer Center ( Site 0047), Albuquerque, New Mexico
  - Presbyterian Rust Jorgensen Cancer ( Site 0073), Rio Rancho, New Mexico
  - Clinical Research Alliance ( Site 0009), Westbury, New York
  - Novant Health Cancer Institute ( Site 0019), Charlotte, North Carolina
  - Novant Health Oncology Specialists ( Site 0074), Winston-Salem, North Carolina
  - TriHealth Cancer Institute-Good Samaritan Hospital ( Site 0020), Cincinnati, Ohio
  - Cancer Care Associates Of York ( Site 0063), York, Pennsylvania
  - JPS Health Network ( Site 0067), Fort Worth, Texas
  - Texas Oncology - Gulf Coast ( Site 8006), Houston, Texas
  - Oncology Consultants P.A. ( Site 0061), Houston, Texas
  - Texas Oncology - Central/South Texas ( Site 8005), McAllen, Texas
  - Mays Cancer Center ( Site 0049), San Antonio, Texas
  - Virginia Oncology Associates (VOA) ( Site 8001), Norfolk, Virginia
  - Shenandoah Oncology ( Site 8004), Winchester, Virginia
  - Northwest Medical Specialties, PLLC ( Site 0062), Tacoma, Washington
  - Circuit Clinical/SSM Health Dean Medical Group ( Site 0039), Madison, Wisconsin
- Argentina (7):
  - Hospital Aleman ( Site 0200), Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0205), Mar del Plata, Buenos Aires
  - Fundación Respirar ( Site 0201), Buenos Aires, Buenos Aires F.D.
  - Centro Privado de RMI Rio Cuarto ( Site 0207), Río Cuarto, Córdoba Province
  - Instituto de Oncología de Rosario ( Site 0208), Rosario, Santa Fe Province
  - Instituto Alexander Fleming ( Site 0202), CABA
  - Hospital Italiano de Córdoba ( Site 0206), Córdoba
- Australia (3):
  - Blacktown Hospital-Blacktown Cancer and Haematology Centre - Medical Oncology ( Site 2300), Blacktown, New South Wales
  - Monash Medical Centre ( Site 2301), Clayton, Victoria
  - The Alfred Hospital ( Site 2305), Melbourne, Victoria
- Liga Norte Riograndense Contra o Câncer ( Site 0301), Natal, Rio Grande do Norte, Brazil
- The Moncton Hospital ( Site 0101), Moncton, New Brunswick, Canada
- Chile (3):
  - Oncovida ( Site 0402), Santiago, Region M. de Santiago
  - Clínica MEDS La Dehesa ( Site 0405), Santiago, Region M. de Santiago
  - CIDO SpA ( Site 0408), Temuco, Región de la Araucanía
- China (16):
  - Anhui Provincial Cancer Hospital ( Site 3140), Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences ( Site 3100), Beijing, Beijing Municipality
  - Peking University People's Hospital. ( Site 3138), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University ( Site 3101), Chongqing, Chongqing Municipality
  - Chongqing Three Gorges Central Hospital's ( Site 3128), Wanzhou, Chongqing Municipality
  - The First Affiliated hospital of Xiamen University ( Site 3120), Fujian, Fujian
  - Sun Yat-Sen University Cancer Center ( Site 3102), Guangzhou, Guangdong
  - Jiangmen Center Hospital ( Site 3132), Jiangmen, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital ( Site 3118), Nanning, Guangxi
  - Jiangsu Province Hospital ( Site 3105), Nanjing, Jiangsu
  - Nanchang People's Hospital ( Site 3124), Nanchang, Jiangxi
  - Affiliated Cancer Hospital of Shandong First Medical University ( Site 3115), Jinan, Shandong
  - Sichuan Cancer Hospital. ( Site 3110), Chengdu, Sichuan
  - West China Hospital of Sichuan University ( Site 3139), Chengdu, Sichuan
  - Sir Run Run Shaw Hospital ( Site 3117), Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province ( Site 3137), Linhai, Zhejiang
- Colombia (5):
  - Instituto de Cancerología-Oncology ( Site 0503), Medellín, Antioquia
  - FUNDACION CTIC CENTRO DE TRATAMIENTO E INVESTIGACION SOBRE CANCER LUIS CARLOS SARMIENTO ANGULO ( Site 0502), Bogotá, Bogota D.C.
  - Instituto Nacional De Cancerologia ( Site 0504), Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS ( Site 0501), Valledupar, Cesar Department
  - IMAT S.A.S ( Site 0500), Montería, Departamento de Córdoba
- France (4):
  - CHRU de Brest ( Site 0904), Brest, Finistere
  - CENTRE LEON BERARD ( Site 0900), Lyon, Rhone
  - Centre de Lutte Contre le Cancer - Centre Henri Becquerel Normandie Rouen ( Site 0901), Rouen, Seine-Maritime
  - Gustave Roussy ( Site 0903), Villejuif, Val-de-Marne
- Greece (4):
  - General Hospital of Athens "Laiko" ( Site 1105), Athens, Attica
  - Aretaieio Hospital ( Site 1103), Athens, Attica
  - University General Hospital of Heraklion ( Site 1102), Heraklion, Irakleio
  - European Interbalkan Medical Center-Oncology Department ( Site 1101), Thessaloniki
- Bacs-Kiskun Varmegyei Oktatokorhaz-Onkoradiologiai Kozpont ( Site 1200), Kecskemét, Bács-Kiskun county, Hungary
- Israel (4):
  - Rambam Health Care Campus ( Site 1401), Haifa
  - Shaare Zedek Medical Center ( Site 1406), Jerusalem
  - Hadassah Medical Center ( Site 1404), Jerusalem
  - Sheba Medical Center ( Site 1400), Ramat Gan
- Italy (5):
  - Azienda Socio Sanitaria Territoriale Papa Giovanni XXIII ( Site 1507), Bergamo, Lombardy
  - Istituto Europeo di Oncologia IRCCS ( Site 1508), Milan, Lombardy
  - Ospedale San Raffaele. ( Site 1502), Milan
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale-S.C. Oncologia Clinica Sperimentale di Senologia ( Site 1506), Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS - Università Cattolica del Sacro Cuore ( Site 1500), Roma
- Japan (14):
  - Nagoya City University Hospital ( Site 3210), Nagoya, Aichi-ken
  - National Hospital Organization Hokkaido Cancer Center ( Site 3215), Sapporo, Hokkaido
  - Kansai Medical University Hospital ( Site 3213), Hirakata, Osaka
  - Kindai University Hospital ( Site 3204), Sakai, Osaka
  - Shizuoka Cancer Center ( Site 3202), Sunto-gun, Shizuoka
  - National Cancer Center Hospital ( Site 3206), Chūō, Tokyo
  - Toranomon Hospital ( Site 3205), Minato, Tokyo
  - Showa Medical University Hospital ( Site 3209), Shinagawa, Tokyo
  - Akita University Hospital ( Site 3207), Akita
  - Chiba Cancer Center ( Site 3203), Chiba
  - National Hospital Organization Kyushu Cancer Center ( Site 3208), Fukuoka
  - Fukushima Medical University Hospital ( Site 3212), Fukushima
  - Hiroshima City Hiroshima Citizens Hospital ( Site 3214), Hiroshima
  - National Hospital Organization Osaka National Hospital ( Site 3201), Osaka
- Poland (2):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie ( Site 1600), Warsaw, Masovian Voivodeship
  - Szpital Kliniczny Ministerstwa Spraw Wewnętrznych i Administracji z Warmińsko-Mazurskim Centrum Onko ( Site 1614), Olsztyn, Warmian-Masurian Voivodeship
- South Korea (6):
  - Seoul National University Bundang Hospital ( Site 2703), Seongnam, Kyonggi-do
  - Gangnam Severance Hospital, Yonsei University Health System ( Site 2701), Gangnam-gu, Seoul
  - Samsung Medical Center ( Site 2704), Gangnam-gu, Seoul
  - Seoul National University Hospital ( Site 2702), Jongno-Gu, Seoul
  - Severance Hospital Yonsei University Health System ( Site 2700), Seoul
  - Asan Medical Center ( Site 2705), Seoul
- Spain (7):
  - Hospital Universitario Marques de Valdecilla ( Site 1825), Santander, Cantabria
  - CHUAC-Complejo Hospitalario Universitario A Coruña ( Site 1820), A Coruña, La Coruna
  - Hospital Clinic de Barcelona ( Site 1821), Barcelona
  - Institut Català d'Oncologia (ICO) - Badalona ( Site 1823), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 1824), Madrid
  - Hospital Clinico San Carlos... ( Site 1822), Madrid
  - Hospital Universitario Virgen de Valme ( Site 1826), Seville
- Taiwan (7):
  - Ditmanson Medical Foundation Chia-Yi Christian Hospital ( Site 2806), Chiayi City, Chiayi
  - Taichung Veterans General Hospital ( Site 2803), Taichung
  - National Cheng Kung University Hospital ( Site 2804), Tainan
  - Chi-Mei Medical Center ( Site 2805), Tainan
  - National Taiwan University Hospital ( Site 2800), Taipei
  - MacKay Memorial Hospital ( Site 2802), Taipei
  - National Taiwan University Cancer Center (NTUCC) ( Site 2801), Taipei
- Bangkok Metropolitan Administration Medical College and Vajira Hospital ( Site 2924), Dusit, Bangkok, Thailand
- Turkey (Türkiye) (6):
  - Hacettepe Universite Hastaneleri ( Site 2100), Ankara
  - Memorial Ankara Hastanesi ( Site 2106), Ankara
  - Ankara Bilkent Şehir Hastanesi ( Site 2105), Ankara
  - Koç Üniversitesi Hastanesi ( Site 2104), Istanbul
  - Mersin Sehir Eğitim ve Araştırma Hastanesi ( Site 2103), Mersin
  - Samsun Medical Park Hastanesi ( Site 2109), Samsun

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — http://www.merckclinicaltrials.com